CLINICAL TRIAL: NCT04512196
Title: Incidence of Surgical Site Infection in Perforated Appendicitis After Peritoneal Lavage With Super-oxidised Solution: A Randomised Double-blind, Placebo-controlled Trial
Brief Title: Surgical Site Infection in Perforated Appendicitis After Peritoneal Lavage With Super-oxidised Solution
Acronym: PLaSSo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Queen Elizabeth, Malaysia (Other Government)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMRR-ID-16-2905-30891
Record Dates: First submitted 2020-05-06; First posted 2020-08-13 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Perforated Appendicitis
Keywords: Perforated Appendicitis; Super-oxidised solution; Surgical site infection; Peritoneal lavage
MeSH Terms: conditions — Appendicitis; Surgical Wound Infection | interventions — superoxidized water; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomised double-blind placebo-controlled parallel-group study. This is a superiority study assessing the effectiveness of the intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study participants, healthcare providers who attend to the participants during the trial (surgeon and nurses), outcome evaluators (surgical doctors and nurses) and data collectors will be blinded to the allocation.
  The sterile study solution (super-oxidised solution) or placebo (normal saline 0.9%) will be stored in a similar storage container and will have the same clear appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super-oxidised Solution (Experimental): Peritoneal lavage with super-oxidised solution of at least 10 cc/kg and wound lavage with super-oxidised solution 1 cc/kg
  Interventions: Drug: Superoxidized Water
- Normal Saline (Placebo Comparator): Peritoneal lavage with normal saline 0.9% of at least 10 cc/kg and wound lavage with normal saline 0.9% 1 cc/kg
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Superoxidized Water — Super-oxidized solution contains hypochlorous acid (HOCl) which exhibits bactericidal activity. These reactive species create an imbalanced osmotic gradient which damages the cell membrane integrity of single celled organisms, and subsequently denaturing its lipid and protein content. Multicellular organisms including host tissue are not susceptible to such changes in osmolarity hence spared from damage.
  Other Names: Hydrocyn Aqua® (Vigilenz MD., Penang, Malaysia); FDA 510(K) Number: K142775
  Arms: Super-oxidised Solution
Drug: Normal Saline — Normal saline contains 0.9% sodium chloride.
  Arms: Normal Saline

SUMMARY:
This study is to evaluate the effectiveness of peritoneal lavage with super-oxidised solution in reducing surgical site infection after open surgery for perforated appendicitis.

DETAILED DESCRIPTION:
Open appendicectomy for perforated appendicitis is associated with significant morbidity from surgical site infection. The standard practice is to perform peritoneal and wound lavage using normal saline solution. The investigators propose the use of superoxidized solution for peritoneal and wound lavage to decrease the incidence of surgical site infection.

Superoxidized solutions contain hypochlorous acid (HOCl) which has bactericidal properties. The reactive oxygen species that is produces damages cell wall membrane of unicellular organisms, however remains safe when in contact with human or animal tissue. It is commonly used for topical treatment of wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age 13 and 70 years
2. Diagnosed with perforated appendicitis intra-operatively
3. Undergo open appendicectomy via Lanz incision

Exclusion Criteria:

1. Surgical technique: Laparoscopic appendicectomy or mid-line laparotomy
2. Patients on steroid treatment and immunosuppressant therapy.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days post surgery
  Number of participants with surgical site infection after open surgery for perforated appendicitis

SECONDARY OUTCOMES:
Inflammatory marker C-reactive protein | 24 and 48 hours post surgery
  Change in serum inflammatory marker C-reactive protein level after open surgery for perforated appendicitis
Post-operative Ileus | From end of surgery till first passage of flatus or bowel opening, whichever comes first, assessed up to 30 days
  Duration of post-operative ileus after open surgery for perforated appendicitis

CONTACTS AND LOCATIONS:
Overall Officials: Hari Sellappan, MB BCh BAO, Principal Investigator — Hospital Queen Elizabeth, Kota Kinabalu, Sabah, Malaysia
Locations (1):
- Hospital Queen Elizabeth, Kota Kinabalu, Sabah, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norman G, Atkinson RA, Smith TA, Rowlands C, Rithalia AD, Crosbie EJ, Dumville JC. Intracavity lavage and wound irrigation for prevention of surgical site infection. Cochrane Database Syst Rev. 2017 Oct 30;10(10):CD012234. doi: 10.1002/14651858.CD012234.pub2. PMID 29083473
- [Background] Kubota A, Goda T, Tsuru T, Yonekura T, Yagi M, Kawahara H, Yoneda A, Tazuke Y, Tani G, Ishii T, Umeda S, Hirano K. Efficacy and safety of strong acid electrolyzed water for peritoneal lavage to prevent surgical site infection in patients with perforated appendicitis. Surg Today. 2015 Jul;45(7):876-9. doi: 10.1007/s00595-014-1050-x. Epub 2014 Nov 13. PMID 25387655
- [Derived] Sellappan H, Alagoo D, Loo C, Vijian K, Sibin R, Chuah JA. Effect of peritoneal and wound lavage with super-oxidized solution on surgical-site infection after open appendicectomy in perforated appendicitis (PLaSSo): randomized clinical trial. BJS Open. 2024 Sep 3;8(5):zrae121. doi: 10.1093/bjsopen/zrae121. PMID 39413050